CLINICAL TRIAL: NCT02560493
Title: Gaming Technology to Encourage Healthy Weight and Activity in Youth
Acronym: GameSquad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 2015-037
Record Dates: First submitted 2015-09-18; First posted 2015-09-25 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Childhood Obesity
Keywords: BMIz; Exergaming; Cardiovascular Disease
MeSH Terms: conditions — Pediatric Obesity; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Condition (No Intervention): Participants randomly assigned to the control condition will be asked to continue their usual physical activity habits and will not interact with the intervention staff.
- Exergaming Condition (Experimental): Participants randomly assigned to the exergaming condition will participate in a 6 month exergaming intervention.
  Interventions: Behavioral: Exergaming Condition

INTERVENTIONS:
Behavioral: Exergaming Condition — Participants are encouraged to meet the MVPA goal of 60 minutes/day, which will be gradually achieved beginning with 10 minutes/day in Week 1 and reaching 60 minutes/day in Week 6. Three hours each week will be devoted to exergame play, following prescribed exergame routines.
  Arms: Exergaming Condition

SUMMARY:
The goal of the proposed randomized controlled trial is to test the efficacy of exergaming (i.e. video gaming that involves physical activity) to reduce adiposity in overweight and obese children.

DETAILED DESCRIPTION:
The GAMESQUAD study is a 6-month, 2-arm randomized controlled trial among 46 overweight/obese children (aged 10 to 12 years) assigned to: 1) 3 hours/week of in-home exergaming or 2) a control group. An innovative aspect is the inclusion of a fitness trainer who will regularly video chat with the participant and virtually monitor gameplay. The study will advance the field by: 1) establishing the efficacy of exergaming to reduce BMIz among overweight and obese children and 2) demonstrating the potential of exergaming to reduce body fat and improve children's cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* BMI percentile > or equal to 85 on the CDC growth chart
* Participating household has a high-speed internet connection
* At least 1 family member or friend who is willing to exergame in the home with the participant for 3 hours/week

Exclusion Criteria:

* Pregnant
* Impairments that prevent normal ambulation
* Previous history, or current symptoms of, cardiovascular disease, musculoskeletal injury, or epileptic seizures

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Staiano, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staiano AE, Beyl RA, Guan W, Hendrick CA, Hsia DS, Newton RL Jr. Home-based exergaming among children with overweight and obesity: a randomized clinical trial. Pediatr Obes. 2018 Nov;13(11):724-733. doi: 10.1111/ijpo.12438. Epub 2018 Jul 20. PMID 30027607

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Condition | Exergaming Condition
Started | 23 | 23
Completed | 22 | 23
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Condition | Exergaming Condition | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (0.8) | 11.3 (0.8) | 11.2 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 15 | 26
  White | 12 | 7 | 19
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46
Body mass index, z-score [Mean (Standard Deviation); unit: z-score.] — The z-score indicates the number of standard deviations away from the mean. A z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean
  z-score. | 2.10 (0.42) | 2.06 (0.46) | 2.08 (0.44)
Fat mass, kg [Mean (Standard Deviation); unit: kg] | 29.3 (7.4) | 30.4 (11.6) | 29.8 (9.6)
Fat mass percentage [Mean (Standard Deviation); unit: percentage of fat mass] | 44.1 (3.4) | 42.0 (5.9) | 43.1 (4.9)
Systolic blood pressure percentile [Mean (Standard Deviation); unit: percentile] | 43.7 (25.9) | 36.4 (11.6) | 40.0 (23.2)
Diastolic blood pressure percentile [Mean (Standard Deviation); unit: percentile] | 63.3 (22.4) | 58.5 (17.8) | 60.9 (20.1)
HDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 51.3 (9.2) | 48.9 (9.1) | 50.1 (9.1)
LDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 99.3 (29.6) | 89.4 (31.2) | 94.4 (30.5)
Moderate-to-vigorous physical activity [Mean (Standard Deviation); unit: minutes/day] — Population: One participant's accelerometry data did not meet standards for completeness (10 hours/day with at least 4 days/week including 1 weekend day).
  minutes/day
    number analyzed (Participants) | 22 | 23 | 45
    (all) | 35.1 (18.3) | 35.0 (17.8) | 35.1 (17.8)
Reported dietary intake [Mean (Standard Deviation); unit: kcal/day] — Population: Some participants did not provide complete data on the dietary recall and were not included in these analyses.
  kcal/day
    number analyzed (Participants) | 22 | 20 | 42
    (all) | 1894.4 (881.2) | 1700.0 (905.4) | 1801.8 (887.3)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Mass Index Z-score (BMIz) Compared to a Control Group
Description: Height and weight will be collected at Screening, Week 0, and Week 24. Standing height will be measured in cm with a Harpenden stadiometer (Holtain Limited, Crymych, UK) with shoes removed while the participant holds breath and an assessor applies light traction to align the participant's head along the Frankfort Horizontal Plane. Weight will be measured in kg with a Michelli GSE 460 scale (G.T. Michelli Co., Baton Rouge, LA) while wearing a hospital gown and undergarments. Measures will be taken twice and recorded to the nearest 0.1 units, with a third if the initial 2 measures are greater than 0.5 units apart. BMIz will be calculated based on the child's age, sex, height, and weight using the 2000 Centers for Disease Control and Prevention (CDC) Growth Charts. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean
Time Frame: Change between Baseline (Week 0) and 6 months (Week 24)
Population: One participant was lost to follow-up.
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Control Condition | Exergaming Condition
Number analyzed (Participants) | 23 | 22
z-score | 0.02 (0.03) | -0.06 (0.03)

2. Secondary Outcome: Changes in Body Fat
Description: A dual energy x-ray absorptiometry (DXA) scan will be completed at Week 0 and Week 24 with a GE iDXA whole-body scanner (GE Medical Systems, Milwaukee, WI) to measure adiposity, including total body fat mass and regional fat mass in the extremities and trunk.
Time Frame: Change between Baseline (Week 0) and 6 months (Week 24)
Population: One participant was lost to follow-up.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Control Condition | Exergaming Condition
Number analyzed (Participants) | 23 | 22
kg | 1.7 (0.5) | 0.8 (0.5)

3. Secondary Outcome: Changes in Systolic Blood Pressure
Description: Resting blood pressure will be assessed at Screening, Week 0, and Week 24 using standard clinical procedures on a standard mercury manometer. The participant's age-, sex-, and height-specific percentile will be calculated.
Time Frame: Change between Baseline (Week 0) and 6 months (Week 24)
Population: One participant was lost to follow-up.
Measure: Least Squares Mean (Standard Error); unit: percentile
Arm/Group | Control Condition | Exergaming Condition
Number analyzed (Participants) | 23 | 22
percentile | 10.9 (5.0) | -5.0 (5.1)

4. Secondary Outcome: Changes in Diastolic Blood Pressure
Description: as for outcome 3
Time Frame: Change between Baseline (Week 0) and 6 months (Week 24)
Population: One participant was lost to follow-up.
Measure: Least Squares Mean (Standard Error); unit: percentile
Arm/Group | Control Condition | Exergaming Condition
Number analyzed (Participants) | 23 | 22
percentile | 8.3 (4.2) | -7.4 (4.3)

5. Secondary Outcome: Changes in Total Cholesterol
Description: A blood sample will be taken at Week 0 and Week 24 by a trained phlebotomist following standard clinic procedures after an 8-hour fast. Serum concentrations of total cholesterol will be assayed on a DXC600 from Trinity.
Time Frame: Change between Baseline (Week 0) and 6 months (Week 24)
Population: One participant was lost to follow-up.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Control Condition | Exergaming Condition
Number analyzed (Participants) | 23 | 22
mg/dL | 6.7 (3.5) | -7.1 (3.5)

6. Secondary Outcome: Changes in Fasting Glucose
Description: A blood sample will be taken at Week 0 and Week 24 by a trained phlebotomist following standard clinic procedures after an 8-hour fast. Serum concentrations of glucose will be obtained from a DXC600 by Beckman Coulter.
Time Frame: Change between Baseline (Week 0) and 6 months (Week 24)
Population: One participant was lost to follow-up.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Control Condition | Exergaming Condition
Number analyzed (Participants) | 23 | 22
mg/dL | 0.4 (1.1) | 0.5 (1.1)

7. Secondary Outcome: Changes in Physical Activity
Description: Physical activity will be assessed with an Actigraph GT3X+ accelerometer (ActiGraph, of Ft. Walton Beach, FL) to determine changes in habitual physical activity outside of the gaming intervention. Participants will wear the accelerometer for two bouts of 7-days following Week 0 baseline clinic visit and Week 24 clinic visit, but not during the gaming intervention.
Time Frame: Change between Baseline (Week 0) and 6 months (Week 24)
Population: Several participants did not meet criteria for complete accelerometry data (at least 4 days of 10 hours/day including 1 weekend day) at both time points.
Measure: Least Squares Mean (Standard Error); unit: minutes/day
Arm/Group | Control Condition | Exergaming Condition
Number analyzed (Participants) | 19 | 16
minutes/day | -7.8 (3.2) | 3.6 (3.4)

8. Secondary Outcome: Changes in Diet
Description: Dietary information will be collected from the participant at Week 0 and Week 24. Healthy diet score will be determined by the NCI Self-administered 24-hour Dietary Recall (ASA24-Kids). This survey is administered on a computer through a web-based program.
Time Frame: Change between Baseline (Week 0) and 6 months (Week 24)
Population: Some participants did not complete the dietary recalls.
Measure: Least Squares Mean (Standard Error); unit: kcal/day
Arm/Group | Control Condition | Exergaming Condition
Number analyzed (Participants) | 22 | 19
kcal/day | 269.5 (200.0) | -297.2 (215.0)

ADVERSE EVENTS:
Arm/Group | Control Condition | Exergaming Condition
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Condition (N=23) | Exergaming Condition (N=23)
Injury during game play (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Bruise to the ankle or wrist

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes